CLINICAL TRIAL: NCT05547243
Title: A Cohort Study to Evaluate Safety and Immunogenicity of COVID-19 mRNA Vaccine, Bivalent (LVRNA021) in Participants Aged 18 Years and Over in China
Brief Title: A Cohort Study of COVID-19 mRNA Vaccine, Bivalent in Participants in China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AIM Vaccine Co., Ltd. (Industry)
Collaborators: Ningbo Rongan Biological Pharmaceutical Co., Ltd. (Industry); The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LVRNA021-IIT-03
Record Dates: First submitted 2022-09-18; First posted 2022-09-21 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2022-09

CONDITIONS: SARS-CoV-2
MeSH Terms: interventions — CVnCoV COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose (Experimental): Two doses were administered by intramuscular injection, 28 days apart
  Interventions: Biological: SARS-CoV-2 mRNA Vaccine, Bivalent Low dose
- High dose (Experimental): Two doses were administered by intramuscular injection, 28 days apart
  Interventions: Biological: SARS-CoV-2 mRNA Vaccine, Bivalent High dose
- Placebo (Placebo Comparator): Two doses were administered by intramuscular injection, 28 days apart
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: SARS-CoV-2 mRNA Vaccine, Bivalent Low dose — 50μg/dose
  Arms: Low dose
Biological: SARS-CoV-2 mRNA Vaccine, Bivalent High dose — 100μg/dose
  Arms: High dose
Drug: Placebo — Saline solution
  Arms: Placebo

SUMMARY:
This is a cohort study to evaluate safety and immunogenicity of COVID-19 mRNA Vaccine, Bivalent (LVRNA021) in participants aged 18 years and over in China

ELIGIBILITY:
Inclusion Criteria:

* Age at the time of first dose of vaccine: adults aged 18-59 years (including boundary values), elderly ≥60 years, both sexes;
* Armpit temperature <37.3℃ on the day of enrollment;
* Based on the medical history and relevant physical examination and laboratory examination results, the investigator clinically determined that the patient was in good health;
* Subjects have independent judgment ability, can read, understand and complete vaccination diary cards, and they participate voluntarily and sign an informed consent form.

Exclusion Criteria:

* The subject has a history of SARS-CoV-2 or SARS infection, or has a history of contact with SARS-CoV-2 infected persons (nucleic acid test positive) or suspected infected persons within 30 days before screening, or living abroad within 30 days before screening history, or a positive SARS-CoV-2 nucleic acid test or a positive SARS-CoV-2 IgM or IgG test before the first dose of vaccine;
* History of allergy to any component of the study vaccine or a history of a severe allergic reaction to the vaccine or drug (including but not limited to anaphylactic shock, anaphylactic laryngeal edema, anaphylactic purpura, thrombocytopenic purpura, or local anaphylactic necrosis [Arthus reaction]);
* Upon questioning, have a history of COVID-19 vaccination, or have received other inactivated vaccines within 14 days before screening, and received live attenuated vaccines within 28 days;
* Patients have a medical history or family history of epilepsy, convulsions, neurological diseases and mental diseases;
* There are contraindications for intramuscular injection, such as: thrombocytopenia that has been diagnosed, any coagulation disorder or receiving anticoagulant treatment, etc.;
* The investigator judges that he is known or suspected of having more serious diseases at the same time, including but not limited to: respiratory diseases (tuberculosis, lung failure, etc.), liver and kidney diseases, cardiovascular diseases (heart failure, severe hypertension, etc.), Malignant tumor, infection or allergic skin disease, HIV infection (test report can be provided), or during the active period of acute infection or chronic disease (within 3 days before vaccination);
* Congenital malformations, developmental disorders, or chronic diseases that the investigator judges are not suitable for participating in this study (such as Downs syndrome, sickle cell anemia or neurological disorders, Guillain-Barre syndrome, etc.), excluding stable diabetes/hypertension );
* Patients with known immunological impairment or low immunological function diagnosed by the hospital before enrollment, or functional asplenia or splenectomy caused by any situation;
* Smokers (≥20 cigarettes per day on average in the past 30 days), alcoholics (≥61 grams of pure alcohol per day on average for men and ≥41 grams of pure alcohol per day for women in the past 30 days) and drug abuse;
* Female: those who have a positive blood pregnancy test, are pregnant, breastfeeding, or have a pregnancy plan within one year; men: whose spouse has a pregnancy plan within one year;
* Patients have participated in other clinical trials (drugs, biological products or devices) within 3 months before the first dose of vaccine, or plan to participate in other clinical trials during the research period;
* Patients received immune enhancement or immunosuppressive therapy within 6 months before the first dose of vaccine (continuous oral or instillation for more than 14 days);
* Patients donated blood ≥400 ml within 28 days before screening, or received whole blood, plasma and immunoglobulin therapy within 6 months before screening;
* Currently receiving research drug treatment to prevent COVID-19;
* Patients are taking antipyretic, analgesic and anti-allergic drugs within 3 days before enrollment;
* The investigator judges that the subjects cannot follow the research procedures, comply with the agreement, or plan to permanently relocate from the area before the end of the research, or plan to leave the local area for a long time during the scheduled visit period;
* The relevant staff involved in this study or their immediate family members (such as spouses, parents, siblings or children);
* According to the investigator's judgment, there are other situations that are not suitable for participating in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 Novel coronavirus S protein antibody (IgG) level | At 28 days after full immunization
The levels of neutralizing antibodies of SARS-CoV-2 anti-Novel coronavirus 2019 (Omicron BA.2, BA.4, BA.5 and Delta strains) true virus | At 28 days after full immunization
The levels of neutralizing antibodies of SARS-CoV-2 anti-Novel coronavirus 2019 (Omicron BA.2, BA.4, BA.5 and Delta strains) pseudovirus | At 28 days after full immunization

SECONDARY OUTCOMES:
Incidence of adverse events | Within 14 days and 28 days after each dose of immunization
Incidence of adverse events associated with the study vaccine | Within 14 days and 28 days after each dose of immunization
Incidence of SAE | Within 28 days, 3 months, 6 months, and 12 months after the first dose of immunization to full immunization
Incidence of AESI | Within 28 days, 3 months, 6 months, and 12 months after the first dose of immunization to full immunization
Incidence of SAE associated with the study vaccine | Within 28 days, 3 months, 6 months, and 12 months after the first dose of immunization to full immunization
Incidence of AESI associated with the study vaccine | Within 28 days, 3 months, 6 months, and 12 months after the first dose of immunization to full immunization
Incidence of grade ≥3 adverse events | Within 28 days after each dose/full dose
Incidence of grade ≥3 adverse events associated with the study vaccine | Within 28 days after each dose/full dose
Statistics of withdrawal from the study due to adverse events | Within 28 days after each dose/full dose
The level of SARS-CoV-2 S protein antibody (IgG) | At 14 days, 3 months, 6 months, and 12 months after full immunization
The positive conversion rate of SARS-CoV-2 S protein antibody | At 14 days, 28 days, 3 months, 6 months, and 12 months after full immunization
True virus neutralizing antibody levels of SARS-CoV-2 (Omicron strain BA.2, BA.4, BA.5, Delta strain) | At 14 days, 3 months, 6 months, and 12 months after full immunization
Pseudovirus neutralizing antibody levels of SARS-CoV-2 (Omicron strain BA.2, BA.4, BA.5, Delta strain) | At 14 days, 3 months, 6 months, and 12 months after full immunization
Positive conversion rates of neutralizing antibodies against true virus of SARS-CoV-2 (Omicron strain BA.2, BA.4, BA.5, Delta strain) | At 14 days, 28 days, 3 months, 6 months, and 12 months after full immunization
Positive conversion rates of neutralizing antibodies against pseudovirus of SARS-CoV-2 (Omicron strain BA.2, BA.4, BA.5, Delta strain) | At 14 days, 28 days, 3 months, 6 months, and 12 months after full immunization
Level of cellular immune response levels (IFN-γ) against Novel coronavirus (2019-nCoV) (ELISPOT) | At 7 days , 14 days , and 28 days after complete immunization
Level of cellular immune response levels ( IL-2) against Novel coronavirus (2019-nCoV) (ELISPOT) | At 7 days , 14 days , and 28 days after complete immunization
Level of cellular immune response levels (IL-4) against Novel coronavirus (2019-nCoV) (ELISPOT) | At 7 days , 14 days , and 28 days after complete immunization
Level of cellular immune response levels (IL-13) against Novel coronavirus (2019-nCoV) (ELISPOT) | At 7 days , 14 days , and 28 days after complete immunization
PBMC transcriptome status at each visit for non-cellular immune subgroup subjects | At 7 days , 14 days , and 28 days after complete immunization

CONTACTS AND LOCATIONS:
Overall Officials: Huan Zhou, Principal Investigator — The First Affiliated Hospital of Bengbu Medical University; Qiang Wu, Principal Investigator — The First Affiliated Hospital of Bengbu Medical University
Locations (1):
- First Affiliated Hospital Bengbu Medical College, Bengbu, Anhui, China